CLINICAL TRIAL: NCT01631994
Title: A Prospective, Single Center, Randomized, Single Blinded Study to Evaluate the Efficacy of Oral Dissolving Metoclopramide Before Video Capsule Endoscopy.
Brief Title: Study to Evaluate the Efficacy of Oral Dissolving Metoclopramide Before Video Capsule Endoscopy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No support to run the study
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: WUH 254286-5
Record Dates: First submitted 2012-06-24; First posted 2012-06-29 (Estimated); Results first posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Gastric Transit Time
Keywords: metoclopramide video capsule endoscopy gastric transit time
MeSH Terms: interventions — Metoclopramide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Dissolving metoclopramide (Experimental): Patient's in this arm will receive the oral dissolving metoclopramide along with the capsule during capsule endoscopy.
  Interventions: Drug: metoclopramide
- control group (No Intervention): This is the control group that will only ingest the capsule during video capsule endoscopy.

INTERVENTIONS:
Drug: metoclopramide — 1 tablet of 10mg of oral dissolving metoclopramide will be taken by patient 45 minutes prior to ingestion of the capsule.
  Arms: Oral Dissolving metoclopramide

SUMMARY:
Summary:

This study investigates the use of oral dissolving metoclopramide during standard video capsule endoscopy. Metoclopramide is a pro -motility agent, that is, this medication helps with movement through the stomach and small bowel. This study will help us determine the effectiveness of oral dissolving metoclopramide on transit time through the stomach and small bowel of the video capsule that is ingested. This study may help with better diagnoses of pathology in the small bowel. Each patient enrolled in the study will either be assigned to a group that only ingests the capsule or the group that receives the oral dissolving metoclopramide plus capsule. Each patient will undergo the same standard procedures and precaution used during standard video capsule endoscopy. The patients that will qualify for the study are patients that are in need of video capsule endoscopy for further imaging of the small bowel. The patients must meet the inclusion criteria provided in the protocol and must not meet any of the exclusion criteria in the protocol. The hypothesis is that the patients that ingest the metoclopramide will have better capsule images and transit time and will allow for enhanced diagnosis of small bowel pathology.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years - 70 years old, male or female, belonging to any race or ethnic origin.
2. Patients necessitating video capsule endoscopy.
3. Patients who are willing and competent to sign an informed consent and to comply with study related visits and procedures.

Exclusion Criteria:

1. Patients below the age of 18 or greater than 70 years old.
2. Pregnant patients
3. Patients with a documented history of Parkinson's Disease or Parkinsonian Symptoms, Tardive Dyskinesia, history of neuroleptic malignant syndrome, history or seizure disorder.
4. Patients who are currently taking antipsychotic medications including typical and atypical antipsychotics.
5. Patients taking other drugs that may cause extrapyramidal reactions.
6. Patients with a history of cirrhosis or congestive heart failure.
7. Patients with a history of depression.
8. Patients with uncontrolled hypertension.
9. Patients with renal impairment, creatinine clearance < 40ml/minute.
10. Patients who have massive gastrointestinal hemorrhage, mechanical obstruction, or perforation.
11. Patients with a known history of pheochromocytoma, as this may precipitate hypertensive crisis.
12. Patients with a known sensitivity or intolerance to metoclopramide.
13. Patients who, in the investigator's opinion, are medically unstable, are unable to give informed consent, or whose risks outweigh the benefits of participating in the study.
14. Vulnerable subjects: Prisoners, persons with decisional incapacity, and any person who are directly involved in the study, including their immediate family members, and anybody who may have any conflict of interest.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Friedel, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was ended early, only 6 patients were enrolled, 2 to the research arm, 4 to the control arm.
Period: Overall Study
Arm/Group | Oral Dissolving Metoclopramide | Control Group
Started | 2 | 4
Completed | 2 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Dissolving Metoclopramide | Control Group | Total
Number analyzed (Participants) | 2 | 4 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (5) | 40 (5) | 40 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Gastric Transit Time
Description: Time for transit through small intestine.
Time Frame: Day 1
Population: No data were collected from the enrolled participants. Study was terminated prior to collection of data.
Arm/Group | Oral Dissolving Metoclopramide | Control Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: No adverse events were collected for this study as it was terminated prior to the collection of data.
Arm/Group | Oral Dissolving Metoclopramide | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No